CLINICAL TRIAL: NCT04034147
Title: The Roots of Metacognitive Failures in Bipolar Disorders: Clinical Determinants of the Discrepancy Between Objective and Subjective Cognition in the Versailles FACE-BD Cohort
Brief Title: Clinical Determinants of the Discrepancy Between Objective and Subjective Cognition in the Versailles FACE-BD Cohort
Acronym: METACOG-BD
Status: Completed | Type: Observational
Sponsor: Versailles Hospital (Other)
Collaborators: Fondation FondaMental (Other)
Responsible Party: Principal Investigator, Dr Paul ROUX, Associated Professor of pqsychiatry, Versailles Hospital
Other Study IDs: Versailles FACE-BD 002
Record Dates: First submitted 2019-07-20; First posted 2019-07-26 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Bipolar Disorder
Keywords: subjective cognition; metacognition; functioning; objective cognition; quality of life; medication adherence
MeSH Terms: conditions — Bipolar Disorder; Medication Adherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Metacognitive abilities have been scarcely investigated in bipolar disorders, with inconsistent results. This may appear somewhat surprising, as metacognitive training is a very promising intervention aiming at improving psychosocial functioning in bipolar disorders. One way to investigate metacognition is to address the discrepancy between objectively measured cognition (through neuropsychological testing) and subjective cognition (through self-reported questionnaire investigating one's perception of cognitive functioning).

Objective and subjective cognition are two fundamental determinants of functioning in bipolar disorder. Objectively-measured cognition is directly associated with performance-based functional capacity but not with self-reported or interview-based functional capacity. In contrast, subjectively-measured cognition is associated with self-reported and interview-based functional capacity, but not performance-based functional capacity.

Associations between subjective cognitive functioning and neuropsychological performances are usually weak, with a moderating effect of manic and depressive symptoms. Manic symptoms are associated with a decrease in cognitive complains, whereas depressive symptoms are associated with an increase in cognitive complaints. Predictors of the discrepancy between objective and subjective cognition in bipolar disorder are still weakly understood. One study reported that the subjective overestimation of cognitive dysfunctioning was positively predicted by more subsyndromal depressive and manic symptoms, hospitalizations, and BD type II. This study also reported that the subjective overestimation of cognitive dysfunctioning was associated with greater socio-occupational difficulties, more perceived stress, and lower quality of life.

However, these previous studies had relatively limited sample sizes (below 150). They also ignored other potential predictors of the discrepancy between objective and subjective cognitions such as psychotic features, impulsiveness, and childhood trauma. Moreover, they also ignored whether this discrepancy was associated with medication adherence.

The present study intends to explore the predictors of the discrepancy between objective and subjective cognition in bipolar disorder in a cross-sectional sample of 387 stable outpatients with bipolar disorders (type 1, type 2, not otherwise specified).

The second objective is to determine whether the discrepancy between objective and subjective cognition in bipolar disorder predicts functioning, quality of life and medication adherence.

DETAILED DESCRIPTION:
Metacognitive abilities have been scarcely investigated in bipolar disorders, with inconsistent results. This may appear somewhat surprising, as metacognitive training is a very promising intervention aiming at improving psychosocial functioning in bipolar disorders. One way to investigate metacognition is to address the discrepancy between objectively measured cognition (through neuropsychological testing) and subjective cognition (through self-reported questionnaire investigating one's perception of cognitive functioning).

Objective and subjective cognition are two fundamental determinants of functioning in bipolar disorder. Objectively-measured cognition is directly associated with performance-based functional capacity but not with self-reported or interview-based functional capacity. In contrast, subjectively-measured cognition is associated with self-reported and interview-based functional capacity, but not performance-based functional capacity.

Associations between subjective cognitive functioning and neuropsychological performances are usually weak, with a moderating effect of manic and depressive symptoms. Manic symptoms are associated with a decrease in cognitive complains, whereas depressive symptoms are associated with an increase in cognitive complaints. Predictors of the discrepancy between objective and subjective cognition in bipolar disorder are still weakly understood. One study reported that the subjective overestimation of cognitive dysfunctioning was positively predicted by more subsyndromal depressive and manic symptoms, hospitalizations, and BD type II. This study also reported that the subjective overestimation of cognitive dysfunctioning was associated with greater socio-occupational difficulties, more perceived stress, and lower quality of life.

However, these previous studies had relatively limited sample sizes (below 150). They also ignored other potential predictors of the discrepancy between objective and subjective cognitions such as psychotic features, impulsiveness, and childhood trauma. Moreover, they also ignored whether this discrepancy was associated with medication adherence.

The present study intends to explore the predictors of the discrepancy between objective and subjective cognition in bipolar disorder in a cross-sectional sample of 387 stable outpatients with bipolar disorders (type 1, type 2, not otherwise specified). All participants were included in the Versailles FACE-BD Cohort and were recruited via the Versailles FondaMental Center of expertise for Bipolar Disorders. BD was diagnosed based on the structured clinical interview that assesses DSM-IV-TR criteria.

Objective cognition was measured with a battery of cognitive tests. Experienced neuropsychologists administered the tests in a fixed order that was the same for every center. Testing lasted a total of 120 min, including 5 to 10-min breaks. The standardized test battery complied with the recommendations issued by the International Society for Bipolar Disorders. It included 11 tests and evaluated the following five cognitive domains:

* processing speed, using the digit symbol coding and symbol search subtests from the Wechsler Adult Intelligence Scale (WAIS) version III, the Trail Making Test (TMT) part A, and the word and the color conditions of the Stroop test
* attention, using the Conners' Continuous Performance Test II (omissions and commissions)
* executive functions, using the colour/word condition of the Stroop test, the TMT part B and verbal fluency (semantic and phonemic conditions)
* verbal memory, using the California Verbal Learning Test (CVLT) immediate recall, short and long delay free recall, and total recognition
* working memory, using the WAIS-III digit span (sum of forward and backward conditions) and the spatial span (forward and backward conditions) subtest from the Wechsler Memory Scale version III

Subjective cognition was measured with item 10 of the Quick Inventory of Depressive Symptomatology-Self-Report-16.

This item focuses over the past 7 days and investigates "Concentration/decision-making:

* 0 There was no change in my usual ability to concentrate or make decisions.
* 1 I occasionally felt indecisive or found that my attention wandered.
* 2 Most of the time, I found it hard to focus or to make decisions.
* 3 I couldn't concentrate well enough to read or I couldn't make even minor decisions"

Predictors of the discrepancy between objective and subjective cognition were:

* type of bipolar disorder
* psychotic features
* age at onset; number of previous mixed, hypomanic, manic, and major depressive episodes; total duration of hospitalizations
* severity of the bipolar disorder with the Clinical Global Impression-Severity
* lithium carbonate, anticonvulsants, antipsychotics, antidepressants, or anxiolytics at the time of testing
* hetero-evaluation of depression with the Montgomery Åsberg Depression Rating Scale
* hetero-evaluation of mania with the Young Mania Rating Scale
* auto-evaluation of the state of anxiety with the state subscale of the State-Trait Anxiety Inventory, form Y-A
* impulsiveness with the Barratt Impulsiveness Scale
* childhood trauma with the Childhood Trauma Questionnaire

The variable predicted by the discrepancy between objective and subjective cognition were:

* the global functioning with the Global Assessment of Functioning scale
* psychosocial functioning in everyday life was assessed with the Functioning Assessment Short Test
* medication adherence with the MEDICATION ADHERENCE RATING SCALE
* quality of life with the EQ-5D

ELIGIBILITY:
Inclusion Criteria:

* bipolar disorder according to DSM IV-R (structured clinical interview)

Exclusion Criteria:

* substance-related disorders in the previous month
* electroconvulsive therapy in the past year
* substantial neurological disorder

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This study included patients recruited into the FACE-BD (FondaMental Advanced Centers of Expertise for Bipolar Disorders) cohort at Versailles Hospital. This registry was set up by the Fondation FondaMental (www.fondation-fondamental. org) which created an infrastructure and provided resources to follow clinical cohorts and comparative-effectiveness research in patients with BD.
  Patients were referred by their general practitioner or by their psychiatrist.
Sampling Method: Non-Probability Sample
Enrollment: 387 (Actual)
Dates: Start 2009-01-01; Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Discrepancy between objective and subjective cognition | one measure per subject, assessed one time at the inclusion
  Sensitivity index scores (rank ordering for subjective performance minus rank ordering for objective performance; minimum -3; maximum 3; higher score indicates greater sensitivity, ie. that subjects reports more subjective complaints compared with their objective neuropsychological performance)

SECONDARY OUTCOMES:
Subjective cognition in individuals without any objective cognitive deficit | one measure per subject, assessed one time at the inclusion
  Subjective cognition measured with item 10 of the Quick Inventory of Depressive Symptomatology-Self-Report-16, minium 0; maximum 3; higher scores indicates worse subjective cognition)
Subjective cognition in individuals with an objective cognitive deficit | one measure per subject, assessed one time at the inclusion
  Subjective cognition measured with item 10 of the Quick Inventory of Depressive Symptomatology-Self-Report-16, minium 0; maximum 3; higher scores indicates worse subjective cognition)

OTHER OUTCOMES:
Global Assessment of Functioning | one measure per subject, assessed one time at the inclusion
  the score on the Global Assessment of Functioning scale (minimum 1; maximum 100; higher scores indicates better functioning)
Psychosocial functioning in everyday life | one measure per subject, assessed one time at the inclusion
  total score on the Functioning Assessment Short Test (lower bound 0 upper bound 72, lower scores indicates better functioning)
Medication adherence | one measure per subject, assessed one time at the inclusion
  Total score on the Medication Adherence Rating Scale (minium 0; maximum 10; lower scores indicates worse adherence)
Quality of Life (domains): EQ-5D-5L | one measure per subject, assessed one time at the inclusion
  Index Value on the EQ-5D-5L (minimum -0.53; maximum 1; higher score indicates better Quality of Life)
Quality of Life (general): visual analogic scale | one measure per subject, assessed one time at the inclusion
  score on the visual analogic scale (minimum 0; maximum 100; higher score indicates better Quality of Life)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Roux, Principal Investigator — Centre Hospitalier de Versailles, Service de psychiatrie de l'adulte
Locations (1):
- Paul ROUX, Le Chesnay, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Haffner P, Quinlivan E, Fiebig J, Sondergeld LM, Strasser ES, Adli M, Moritz S, Stamm TJ. Improving functional outcome in bipolar disorder: A pilot study on metacognitive training. Clin Psychol Psychother. 2018 Jan;25(1):50-58. doi: 10.1002/cpp.2124. Epub 2017 Aug 30. PMID 28857347
- [Background] Lin X, Lu D, Huang Z, Chen W, Luo X, Zhu Y. The associations between subjective and objective cognitive functioning across manic or hypomanic, depressed, and euthymic states in Chinese bipolar patients. J Affect Disord. 2019 Apr 15;249:73-81. doi: 10.1016/j.jad.2019.02.025. Epub 2019 Feb 6. PMID 30763798
- [Background] Miskowiak KW, Petersen JZ, Ott CV, Knorr U, Kessing LV, Gallagher P, Robinson L. Predictors of the discrepancy between objective and subjective cognition in bipolar disorder: a novel methodology. Acta Psychiatr Scand. 2016 Dec;134(6):511-521. doi: 10.1111/acps.12649. Epub 2016 Sep 20. PMID 27644707
- [Background] Ott C, Mine H, Petersen JZ, Miskowiak K. Relation between functional and cognitive impairments in remitted patients with bipolar disorder and suggestions for trials targeting cognition: An exploratory study. J Affect Disord. 2019 Oct 1;257:382-389. doi: 10.1016/j.jad.2019.07.030. Epub 2019 Jul 5. PMID 31302528
- [Background] Rush AJ, Trivedi MH, Ibrahim HM, Carmody TJ, Arnow B, Klein DN, Markowitz JC, Ninan PT, Kornstein S, Manber R, Thase ME, Kocsis JH, Keller MB. The 16-Item Quick Inventory of Depressive Symptomatology (QIDS), clinician rating (QIDS-C), and self-report (QIDS-SR): a psychometric evaluation in patients with chronic major depression. Biol Psychiatry. 2003 Sep 1;54(5):573-83. doi: 10.1016/s0006-3223(02)01866-8. PMID 12946886
- [Background] Van Camp L, Sabbe BGC, Oldenburg JFE. Metacognitive functioning in bipolar disorder versus controls and its correlations with neurocognitive functioning in a cross-sectional design. Compr Psychiatry. 2019 Jul;92:7-12. doi: 10.1016/j.comppsych.2019.06.001. Epub 2019 Jun 6. PMID 31202082
- [Background] Yatham LN, Torres IJ, Malhi GS, Frangou S, Glahn DC, Bearden CE, Burdick KE, Martinez-Aran A, Dittmann S, Goldberg JF, Ozerdem A, Aydemir O, Chengappa KN. The International Society for Bipolar Disorders-Battery for Assessment of Neurocognition (ISBD-BANC). Bipolar Disord. 2010 Jun;12(4):351-63. doi: 10.1111/j.1399-5618.2010.00830.x. PMID 20636632